CLINICAL TRIAL: NCT03142256
Title: A Pilot Prospective Cohort Evaluation of Uptake and Adherence to PrEP in Young South African Women
Brief Title: 3Ps for Prevention Study (Perception, Partners, Pills)
Acronym: 3P
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Desmond Tutu HIV Centre (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); National Institute of Mental Health (NIMH) (NIH); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3P
Record Dates: First submitted 2017-03-03; First posted 2017-05-05 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Adherence
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Incentivised - Conditional Cash Transfer (Active Comparator): Cash incentive for good drug levels assed by Dried Blood Spot
  Interventions: Behavioral: Incentivised - Conditional Cash Transfer; Drug: Truvada 200Mg-300Mg Tablet
- No incentive (No Intervention): Truvada 200Mg-300Mg Tablet

INTERVENTIONS:
Behavioral: Incentivised - Conditional Cash Transfer — Participant will be randomized to receive a cash transfer conditional on drug levels at months 1, 2, and 3 versus no cash transfer
  Other Names: Truvada 200Mg-300Mg Tablet
  Arms: Incentivised - Conditional Cash Transfer
Drug: Truvada 200Mg-300Mg Tablet — Both study arms will be offered Truvada as PrEP. Only one arm will be randomized to the conditional cash transfer.
  Other Names: Incentivised - Conditional Cash Transfer
  Arms: Incentivised - Conditional Cash Transfer

SUMMARY:
This study has two phases. It will be conducted in one site in CT only. Phase I is to enumerate interest in PrEP uptake among young South African women exposed to a culturally-appropriate social marketing campaign. This enumeration will also serve as a recruitment strategy for a cohort with open-label PrEP access in Phase II. The cohort will assess PrEP acceptability and adherence among 200 HIV-uninfected young women who are offered open-label daily oral PrEP and randomized to receive or not receive a short term cash incentive conditional on study drug adherence.

DETAILED DESCRIPTION:
3P for Prevention Study (Perception, Partners, Pills) Synopsis A Pilot Prospective Cohort Evaluation of Uptake and Adherence to PrEP in Young South African Women Background: Despite the wide scale implementation of antiretroviral treatment as prevention and HIV testing, the HIV incidence among young South African women remains unacceptably high, with recent HIV Prevention trials in the Western Cape documenting an incidence as high as 5-6% per year.

In collaboration with others, we conducted formative research in Masiphumelele about the content and format of a communication campaign with clear and compelling messages about PrEP that could increase PrEP demand among young at-risk women in the community context. McCann is currently developing a social marketing campaign about oral PrEP, based on these results. This campaign will be used during the recruitment of this cohort. In addition to understanding what will initially attract women to PrEP, for those women who choose to take PrEP, there is a need to understand adherence support interventions that are scalable and sustainable. Drawing on behavioural economics theories, recent trials of young African women have shown that financial incentives can improve health behaviour.

This study has two phases. It will be conducted in one site in CT only. Phase I is to enumerate interest in PrEP uptake among young South African women exposed to a culturally-appropriate social marketing campaign. This enumeration will also serve as a recruitment strategy for a cohort with open-label PrEP access in Phase II. The cohort will assess PrEP acceptability and adherence among 200 HIV-uninfected young women who are offered open-label daily oral PrEP and randomized to receive or not receive a short term cash incentive conditional on study drug adherence.

Design:

Using the results of the 2016 census, recruitment staff will identify the homes of up to 1000 young women currently between the ages of 16-25. Up to 800 women will be shown a video explaining oral PrEP and take a short survey before and after the video. The survey questions will include demographics, sexual relationships, risk taking, and knowledge and opinions about PrEP. The remaining 200 women will not be shown the video but will be asked the survey questions to serve as a comparison group to evaluate the effect of the PrEP video on initial interest in PrEP. Young women who are interested in learning more about oral PrEP will be referred to community education sessions. We will document the number of women who are interested in learning more about PrEP and the number of attendees at the educational sessions.

Young women interested in taking oral PrEP, regardless if they learned about it through the household video recruitment or community educational sessions, will be referred to the study site to determine if they are eligible for the Phase II cohort. Women who consent to be screened will have their survey data linked to their participant identification number. By linking the data from the surveys conducted during household recruitment and community education events with screening and enrolment, we will be able to assess the PrEP demand and characteristics of women who seek additional information about PrEP, and the subset of those who accept and initiate PrEP.

Phase II: Cohort Study of PrEP in Young Women Objectives I. Primary Objective a. To assess the effect of an incentive provided at months 2, 3, and 6 and conditioned on young women's PrEP adherence, measured by PrEP drug levels at 1, 2, and 3 months after initiating PrEP II and the primary outcome is measured by tenofovir drug levels ≥700 fmol/punch at Month 3 and secondary outcomes at Months 6 and 12.Secondary Objective

1. To assess the durability of the effect of an incentive conditioned on young women's PrEP adherence, as measured by tenofovir drug levels at Months 6, 9, and 12.
2. To explore factors, including knowledge of current partner HIV status, that influence young women's PrEP initiation and adherence over 12 months
3. To assess the social benefits and harms associated with PrEP use III. Exploratory Objective

a. To assess HIV incidence among PrEP users, and PrEP adherence and resistance among women who seroconvert Study Population 200 sexually active HIV-1 uninfected young women 16-25 years old in Masiphumelele township, Cape Town, South Africa who are not currently enrolled in any other research studies and have not previously participated in an oral PrEP study.

Inclusion Criteria Female at birth; HIV uninfected at screening and enrolment; Age 16-25 years old at screening, inclusive; Per participant report, sexually active, defined as having vaginal or anal intercourse with a male partner at least once in the month prior to enrolment; Willing and able to provide informed consent; Able and willing to provide adequate locator information; Tanner stage ≥ 3.

Exclusion Criteria Young women who have met any of the following criteria will be excluded from this study: A positive HIV test at enrolment; Renal dysfunction (Creatinine Clearance <60 mL/min, Cockroft-Gault equation); Previous participation in an oral PrEP study.

Design Screening and Enrollment At the screening visit, women who meet the inclusion and exclusion criteria will be consented. Women will be randomized to receive a small monetary incentive conditioned on PrEP adherence in addition to real time feedback about adherence, using dried blood spots (DBS) to assess PrEP drug levels verses real time feedback and supportive adherence counselling.

Follow-up Visits At all follow-up visits, women will have HIV-1 testing, STI surveillance, partnership characteristics, behavioral data, and medical history data collected. At Months 6 and 12, women will have diagnostic testing for STIs and creatinine testing.

All participants who accept PrEP will receive adherence counselling at each visit and a DBS collected for storage. All women will have DBS PrEP drug level concentration testing at Months 1, 2,3,6 & 12. For Month 1,2 & 3 women who are randomized to the incentive arm will receive real time feedback about their intracellular drug levels and counseling. Women who have a detectable DBS PrEP drug level will receive the cash incentive and will be counselled on adherence to PrEP in order to get optimal HIV protection against HIV and explore barriers to taking PrEP. Women who have an undetectable PrEP drug level at Month 1, 2, or 3 in the incentive arm will receive adherence counseling to take PrEP but they will not receive the incentive for that visit. Women who are not randomized to receive the incentive will receive real time feedback about their intracellular drug levels and supportive adherence counseling as detailed above.

Seroconversion Participants will have rapid HIV testing per national algorithm at each study visit prior to administration of PrEP. Any participant who is confirmed to have acquired HIV during the study will permanently discontinue PrEP and will be transitioned to a local HIV care clinic as per DTHF SOP.

Withdrawal Participants may voluntarily decide to withdraw from the study for any reason at any time. The site investigator may also withdraw participants from the study to protect their safety.

Qualitative Interviews We will randomly select up to 24 women to participate in qualitative interviews exploring women's decision making about PrEP initiation and continuation, barriers and facilitators to PrEP adherence, and whether they disclosed their PrEP use with family members, peers, and their partner(s).

Involvement of minor women, particularly young women, continue to bear a disproportionate burden of HIV in South Africa. The application of novel biomedical prevention tools may be able to prevent a substantial number of HIV infections among young women. We have had indications that youth are willing to engage in more information and community participation around these topics.

ELIGIBILITY:
Inclusion Criteria:

* Female at birth
* HIV uninfected at screening and enrollment
* Age 16-25 years old at screening, inclusive
* Per participant report, sexually active, defined as having vaginal or anal intercourse with a male partner at least once in the month prior to screening
* Willing and able to provide informed consent
* Able and willing to provide adequate locator information

Exclusion Criteria:

* Not planning to be in the area for periods longer than a month in the first three months and longer than 3 months from Month 3 - 12
* A positive HIV test at Enrollment, even if subsequent testing indicates that the person is HIV-1 uninfected
* Renal dysfunction (Creatinine Clearance <60 mL/min, Cockroft Gault equation)
* Previous participation in an oral PrEP study

Ages: 16 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Drug adherence | 3 months
  200 women measuring cash incentive for drug adherence with half the Cohort

CONTACTS AND LOCATIONS:
Locations (2):
- South Africa (2):
  - Desmond Tutu HIV Foundation, Cape Town, Western Cape
  - Desmond Tutu HIV Centre, Cape Town

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Celum CL, Gill K, Morton JF, Stein G, Myers L, Thomas KK, McConnell M, van der Straten A, Baeten JM, Duyver M, Mendel E, Naidoo K, Dallimore J, Wiesner L, Bekker LG. Incentives conditioned on tenofovir levels to support PrEP adherence among young South African women: a randomized trial. J Int AIDS Soc. 2020 Nov;23(11):e25636. doi: 10.1002/jia2.25636. PMID 33247553
- [Derived] Morton JF, Myers L, Gill K, Bekker LG, Stein G, Thomas KK, Duyver M, van der Straten A, McConnell M, Aunger R, Curtis V, de Witt Huberts J, Van Damme L, Baeten JM, Celum C. Evaluation of a behavior-centered design strategy for creating demand for oral PrEP among young women in Cape Town, South Africa. Gates Open Res. 2020 Jul 3;4:29. doi: 10.12688/gatesopenres.13103.2. eCollection 2020. PMID 32411946